CLINICAL TRIAL: NCT02951598
Title: Longitudinal Cohort Study of Resource Use and Cost of Mild Cognitive Impairment and Mild Dementia Due to Alzheimer's Disease in the United States (GERAS-US)
Brief Title: A Study of Health Care Use and Costs in Participants With Early Stage Alzheimer's Disease (AD)
Acronym: GERAS-US
Status: Active, not recruiting | Type: Observational
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Other Study IDs: 16466; H8A-US-B004 (Other: Eli Lilly and Company)
Record Dates: First submitted 2016-10-28; First posted 2016-11-01 (Estimated); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Alzheimer Disease; Mild Cognitive Impairment
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- MCI (Amyloid Positive): Participants with mild cognitive impairment (MCI) due to AD who tested amyloid positive were observed for up to 36 months. No therapeutic investigational drug intended to treat AD was administered.
  Interventions: Drug: Florbetapir F 18 PET Scan
- Mild AD Dementia (Amyloid Positive): Participants with mild AD dementia who tested amyloid positive were observed for up to 36 months. No therapeutic investigational drug intended to treat AD was administered.
  Interventions: Drug: Florbetapir F 18 PET Scan
- MCI (Amyloid Negative): Participants with MCI who tested amyloid negative. These participants were not eligible to participate in the 36 month prospective portion of the study.
  Interventions: Drug: Florbetapir F 18 PET Scan
- Mild Dementia (Amyloid Negative): Participants with mild dementia who tested amyloid negative. These participants were not eligible to participate in the 36 month prospective portion of the study.
  Interventions: Drug: Florbetapir F 18 PET Scan

INTERVENTIONS:
Drug: Florbetapir F 18 PET Scan — Florbetapir F 18 positron emission tomography (PET) scan performed at baseline to confirm amyloid status. Participants who previously tested amyloid positive were exempt. No therapeutic investigational drug(s) intended to treat AD will be administered.
  Other Names: LY3078786

SUMMARY:
The purpose of this study is to learn about health care use, costs, and clinical outcomes over time for amyloid positive participants with early stages of AD in the United States. This study is for research purposes only, and is not intended to treat any medical condition. No study therapy(ies) for AD will be administered.

ELIGIBILITY:
Inclusion Criteria:

* Presents within normal course of outpatient care for whom the physician deems to meet clinical criteria for MCI due to AD or mild AD dementia.
* Fully informed written consent of the participant (or his/her legal representative).
* Study partner who has frequent contact with the participant is willing to accompany the participant at the study observations.
* Fully informed written consent of the study partner; this person must be willing to serve as study partner for at least 6 months of the year.
* Able to communicate in English and/or US Spanish.
* Able to provide evidence of amyloid testing.
* Has an Mini-Mental State Examination (MMSE) score of 20 or greater.

Exclusion Criteria:

* Are currently enrolled in any other clinical trial involving an investigational product or any other type of medical research judged not to be scientifically or medically compatible with this study at baseline.
* Are investigator site personnel directly affiliated with this study and/or their immediate families. Immediate family is defined as a spouse, parent, child, or sibling, whether biological or legally adopted.
* Lack of evidence of amyloid positivity through pre-study test. Note: After baseline assessment, participants with amyloid negativity identified as part of the study will not continue in post-baseline assessments.
* Are Lilly employees or are employees of any third-party organization (TPO) involved in study who require exclusion of their employees.

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1400 (Estimated)
Dates: Start 2016-10-29 (Actual); Primary Completion 2021-01-30 (Actual); Study Completion 2026-04-28 (Estimated)

PRIMARY OUTCOMES:
Mean Economic Cost Associated with Amyloid Positive AD | Baseline through Study Completion (36 Months)

SECONDARY OUTCOMES:
Healthcare Resource Use by AD Cohort | Baseline through Study Completion (36 Months)
Mean Economic Cost by AD Cohort | Baseline through 24 Months
Bath Assessment of Subjective Quality of Life in Dementia (BASQID) | Baseline, End of Study (36 Months)
Mini-Mental State Examination (MMSE) | Baseline, End of Study (36 Months)
Alzheimer's Disease Assessment Scale - Cognitive Subscale (ADAS-Cog14) | Baseline, End of Study (36 Months)
Neuropsychiatric Inventory (NPI) | Baseline, End of Study (36 Months)
Functional Activities Questionnaire (FAQ) | Baseline, End of Study (36 Months)
Cognitive Function Inventory (CFI) | Baseline, End of Study (36 Months)
Zarit Burden Interview (ZBI) | Baseline, End of Study (36 Months)
Percentage of Participants with a Change in Living Situation | 36 Months
Time to Transition Across Stages of AD | Baseline through Study Completion (36 Months)
Desire to Institutionalize Scale (DTI) | Baseline through Study Completion (36 Months)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (76):
- United States (76):
  - California Pharmaceutical Research Institute, Anaheim, California
  - Advanced Research Center, Anaheim, California
  - Sun Valley Research Center, Imperial, California
  - Global Clinical Trials, Irvine, California
  - Irvine Clinical Research Center, Irvine, California
  - Alliance Research Centers, Laguna Hills, California
  - Pacific Clinical Studies, Inc, Los Alamitos, California
  - California Neurological Services, Inc., Panorama City, California
  - Havana Research Institute, Pasadena, California
  - Clinical Innovations, Inc., Riverside, California
  - Breakthrough Clinical Trials, San Bernardino, California
  - HB Clinical Trials, Santa Ana, California
  - Ventura Clinical Trials, Ventura, California
  - Colorado Neurological Institute, Englewood, Colorado
  - Coastal Connecticut Research, LLC, New London, Connecticut
  - JEM Research Institute, Atlantis, Florida
  - Visionary Investigators Network, Aventura, Florida
  - Research Alliance, Clearwater, Florida
  - Clinical Research of South Florida, Coral Gables, Florida
  - Infinite Clinical Research, Doral, Florida
  - International Research Partners, LLC., Doral, Florida
  - Sarkis Clinical Trials, Gainesville, Florida
  - Indago Research & Health Center, Inc., Hialeah, Florida
  - New Life Medical Research Center, Inc, Hialeah, Florida
  - Galiz Research, Hialeah, Florida
  - South Florida Clinical Trials, Hialeah, Florida
  - Van Buren Medical, Hollywood, Florida
  - Clinical Research of Homestead, Homestead, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Universal Neurological Care, Jacksonville, Florida
  - Sunrise Medical Research, Lauderdale Lakes, Florida
  - Biomed Research Institute, Miami, Florida
  - Miami Jewish Health Systems, Miami, Florida
  - Florida International Research Center, Miami, Florida
  - The Neurology Research Group, LLC, Miami, Florida
  - L&C Professional Medical Research Institute, Miami, Florida
  - Genoma Research Group, Inc., Miami, Florida
  - Empire Clinical Research, Miami Lakes, Florida
  - Medical Research Group of Central Florida, Orange City, Florida
  - Combined Research Orlando Phase I-IV LLC, Orlando, Florida
  - Suncoast Neuroscience Associates, St. Petersburg, Florida
  - Stedman Clinical Trials, Tampa, Florida
  - Asclepes Research Centers Florida, Weeki Wachee, Florida
  - Doctors Clinical Research, Atlanta, Georgia
  - American Health Network, Franklin, Indiana
  - American Research, LLC, Jeffersonville, Indiana
  - Heartland Research Associates, Newton, Kansas
  - Baptist Health Medical Group, Lexington, Kentucky
  - NeuroMedical Clinic of Central Louisiana, Alexandria, Louisiana
  - St. Agnes Medical Group, Catonsville, Maryland
  - Hattiesburg Clinic, Hattiesburg, Mississippi
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Psych Care Consultants Research, St Louis, Missouri
  - Pyramid Clinical Research, Monroe, New Jersey
  - Healthwise Medical Associates, PC, Brooklyn, New York
  - Integrative Clinical Trials, LLC, Brooklyn, New York
  - Adirondack Medical Center, Lake Placid, New York
  - Mid Hudson Medical Research, PLLC, New Windsor, New York
  - Onsite Clinical Solutions, LLC, Charlotte, North Carolina
  - Alzheimer's Memory Center, Charlotte, North Carolina
  - Coastal Carolina Healthcare, P.A., New Bern, North Carolina
  - Dayton Center for Neurological Disorders, Centerville, Ohio
  - Christ Hospital, Cincinnati, Ohio
  - Family Practice Center of Wooster, Wooster, Ohio
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Wesley Neurology Clinic, Cordova, Tennessee
  - Clinical Research Solutions, P.C., Knoxville, Tennessee
  - Lakeside Life Center, Carrollton, Texas
  - Univ Of Texas Southwestern at Dallas Childrens Med Ctr, Dallas, Texas
  - The Clinical Research Group, Frisco, Texas
  - Dallas Clinical Research, Greenville, Texas
  - Highlands Medical Associates, P.A., Highlands, Texas
  - University Hills Clinical Research, Irving, Texas
  - North Pointe Psychiatry, Lewisville, Texas
  - Premier Clinical Research, Spokane, Washington

IPD SHARING:
Plan to Share IPD: Yes
Lilly provides access to the individual patient data from studies on approved medicines and indications as defined by the sponsor specific information on ClinicalStudyDataRequest.com.
  This access is provided in a timely fashion after the primary publication is accepted. Researchers need to have an approved research proposal submitted through ClinicalStudyDataRequest.com. Access to the data will be provided in a secure data sharing environment after signing a data sharing agreement.

REFERENCES:
- [Derived] Robinson RL, Rentz DM, Bruemmer V, Scott Andrews J, Zagar A, Kim Y, Schwartz RL, Ye W, Fillit HM. Observation of Patient and Caregiver Burden Associated with Early Alzheimer's Disease in the United States: Design and Baseline Findings of the GERAS-US Cohort Study1. J Alzheimers Dis. 2019;72(1):279-292. doi: 10.3233/JAD-190430. PMID 31561360